CLINICAL TRIAL: NCT06034509
Title: Cognitive and Vascular Functioning Following TBI
Status: Recruiting | Type: Observational
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: WRNMMC-2022-0409; W81XWH-22-2 (Other Grant/Funding Number: CDMRP)
Record Dates: First submitted 2023-04-17; First posted 2023-09-13 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-07

CONDITIONS: Traumatic Brain Injury; Cognitive Decline; Vascular Dementia
Keywords: Traumatic Brain Injury; Cognitive Decline; Vascular Dementia; Blood Biomarkers; Cerebrovascular Reactivity; Military
MeSH Terms: conditions — Brain Injuries, Traumatic; Cognitive Dysfunction; Dementia, Vascular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood serum and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- TBI Group: Participants in this group will have been identified as sustaining a traumatic brain injury (mild, moderate, severe, or penetrating).
  Interventions: Other: No intervention. This is an observational study.
- High-blast exposed control group: Participants in this group will have no history of traumatic brain injury AND will have a lifetime history of greater than 10 blast exposures.
  Interventions: Other: No intervention. This is an observational study.
- Low-blast exposed control group: Participants in this group will have no history of traumatic brain injury AND will have a lifetime history of less than 10 blast exposures.
  Interventions: Other: No intervention. This is an observational study.

INTERVENTIONS:
Other: No intervention. This is an observational study. — There are no interventions being tested in the Cognitive and Vascular Functioning Following TBI study.

SUMMARY:
This observational study will examine the association of chronic traumatic cerebrovascular injury and cardiovascular risk factors with TBI-related cognitive impairment and vascular dementia. Cerebrovascular, inflammatory, and neurodegenerative blood biomarkers as well as clinical and neuroimaging data

DETAILED DESCRIPTION:
The investigators will enroll 300 Service Members (SMs) and Veterans who participated in the National Intrepid Center of Excellence (NICoE) intensive outpatient program or Defense and Veterans Brain Injury Center/Traumatic Brain Injury Center of Excellence (DVBIC/TBICoE) 15-Year TBI Natural History of TBI Study (NatHx) at least three years prior to the present evaluation and provided prior blood specimens stored for analysis. Following informed consent, participants will undergo semi-structured interviews assessing posttraumatic stress disorder (PTSD) and updated lifetime TBI history, neurological examination, neuropsychological testing, structural Magnetic Resonance Imaging (MRI) T1, T2, fluid attenuated inversion recovery (FLAIR), diffuse tensor imaging (DTI), as well as novel imaging techniques to assess imaging biomarkers of traumatic cerebrovascular injury (TCVI): 1) functional MRI (fMRI)-Blood Oxygen Level Dependent (BOLD) with hypercapnia challenge to measure cerebrovascular reactivity (CVR); and 2) Dynamic Contrast Enhanced-MRI to assess blood brain barrier integrity, and an additional research blood draw [apolipoprotein E (APOE) genotype; plasma biomarkers including vascular (e.g., vascular endothelial growth factor, von Willebrand Factor, cholesterol, homocysteine), inflammatory (e.g., high sensitivity c-reactive protein, interleukin-6 (IL-6), chitinase-3-like protein 1 (YKL-40)), and neuronal degeneration (e.g., neurofilament light, phosphorylated tau, brain-derived neurotrophic factor, beta amyloid proteins)]. A medical record review will be conducted specifically for current and past history of cerebrovascular risk factors (e.g., hypertension, diabetes, tobacco use) and psychological conditions (e.g., PTSD, depression). The project will also leverage previously collected data, comparing participants' symptoms, cognitive performance, imaging, and, blood biomarkers to those previously collected through the NICoE, 15-Year study and/or the DOD serum repository, with data from at least two time points on all individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Active duty uniformed SM or Veteran who is currently eligible for treatment at WRNMMC (i.e., Defense Enrollment Eligibility Reporting System (DEERS)-eligible).
2. Ability to read, write, and speak English.
3. Ability to provide informed consent.
4. NICoE Intensive Outpatient Program (IOP) or NatHx Study comprehensive evaluation ≥3 years prior to current evaluation with valid neuropsychological test results.
5. Consent to allow access to prior research data collected through the NICoE TBI Neuroimaging Core Project or NatHx Study and consent to allow access to at least 1 prior blood specimen previously collected through these studies or the DoD Serum Biorepository.

Additional TBI Inclusion Criteria

1. History of at least one mild, moderate, severe, or penetrating TBI > 3 years prior to enrollment. TBI will be diagnosed if any one of the following criteria immediately after the injury is met and attributed to the brain injury, rather than environmental/psychological/other injury factors (DoD-VA criteria246):

1. Loss of consciousness (LOC) or post-traumatic amnesia (PTA)
2. Alteration of consciousness (AOC)
3. Evidence of neurologic dysfunction
4. TBI-related abnormality on structural neuroimaging (either CT or MRI). Additional Healthy Control Criteria

   1. History of military deployment.
   2. Low history of blast exposure (i.e., <10 blasts) Additional Blast Control Criteria

   <!-- -->

   1. History of significant blast exposure (i.e., exposure to ≥ 10 blasts)

Exclusion Criteria:

1. Disabling neurologic or psychological disorders such as autism, cerebral palsy, developmental disorder, stroke, brain tumor, multiple sclerosis, meningitis, encephalitis, brain abscess, vascular malformation, pre-injury epilepsy, schizophrenia, bipolar disorder, personality disorder
2. Diabetes mellitus requiring drug treatment
3. Hypertension requiring more than 1 antihypertensive drug to control BP
4. History of myocardial infarction or other systemic vasculopathies
5. Dementia diagnosis at initial NICoE/NatHx Study assessment

Ages: 18 Years to 74 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male and female active duty service members or DEERS-eligible veterans at least 18 years of age who have participated in the NICoE Intensive Outpatient Program or 15 Year Natural History Study will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Panel of blood biomarkers | 3 years
  A panel of blood biomarkers including vascular (e.g., vascular endothelial growth factor, von Willebrand Factor, cholesterol, lipoproteins, homocysteine, fibrinogen, hemoglobin A1C), inflammatory (e.g., high sensitivity c-reactive protein, Tumor Necrosis Factor-alpha, IL-6, IL-12p70, YKL-40), and neuronal degeneration (e.g., neurofilament light, Glial Fibrillary Acidic Protein, phosphorylated tau, Clusterin, brain-derived neurotrophic factor, beta amyloid proteins) will be compared between TBI groups. One-way ANOVAs will be run with TBI severity as the independent variable and each individual blood biomarker (measured in pg/mL) as the dependent variable. Spearman's rank order correlations will evaluate the relationship between blood biomarkers, number of TBIs, and TBI severity.
Cognitive Performance- Overall Test Battery Mean | 3 years
  Neurocognitive data will be corrected for age, gender, education, and race, as available. An overall test battery mean (OTBM) T-score will be calculated as the average of seven cognitive domain T-scores (attention/processing speed, working memory, executive functioning, learning/immediate memory, delayed memory, language, perceptual reasoning). Each biomarker will be correlated with the OTBM using Spearman's rank order correlations. Cognitive domain T-scores will also be evaluated to understand which are driving changes in the OTBM. All scores will be evaluated as T-scores (mean=50, SD=10, min=0, max=100), for which higher scores indicate higher cognitive performance. Multivariable logistic regression will be used to evaluate the relationship between TBI number, TBI severity, blood biomarkers and normal cognition vs. mild cognitive impairment (MCI).

SECONDARY OUTCOMES:
Change in panel of blood biomarkers over time | 3 years
  Linear mixed effect (LME) models will be fit to the analysis dataset which use the panel of blood biomarkers as the response variables and investigate TBI severity, number of TBI events, and time. The panel of blood biomarkers will include vascular (e.g., vascular endothelial growth factor, von Willebrand Factor, cholesterol, lipoproteins, homocysteine, fibrinogen, hemoglobin A1C), inflammatory (e.g., high sensitivity c-reactive protein, Tumor Necrosis Factor-alpha, IL-6, IL-12p70, YKL-40), and neuronal degeneration (e.g., neurofilament light, Glial Fibrillary Acidic Protein, phosphorylated tau, Clusterin, brain-derived neurotrophic factor, beta amyloid proteins) biomarkers, all measured in pg/mL.
Change in overall test battery mean over time | 3 years
  The investigators will fit a cross-sectional multivariable regression model to the data with the response variable being the change (Time 3 - Time 2) in the OTBM T-score (mean=50, SD=10, min=0, max=100). Individual cognitive domain composite T-scores will also be evaluated to understand the main components driving change in the OTBM.
Change in brain volume over time | 3 years
  The investigators will fit a cross-sectional multivariable regression model to the data with the response variable being the change (Time 3 - Time 2) in total brain volume [milliliters (mL)].
Change in white matter lesions over time | 3 years
  The investigators will fit a cross-sectional multivariable regression model to the data with the response variable being the change (Time 3 - Time 2) in total and total number of white matter lesions.
Cerebrovascular Reactivity | 3 years
  Linear regression models will be run with the difference score in each vascular blood biomarker from the initial visit to the current study visit as the independent variable and global CVR (%S/mmHG) - (assessed during the current visit only) as the dependent variable.
DCE-MRI | 3 years
  Linear regression models will be run with the difference score in each vascular blood biomarker from the initial visit to the current study visit as the independent variable and overall blood brain barrier function (assessed during the current visit only as the percentage of brain volume with suprathreshold voxels) as the dependent variable.

CONTACTS AND LOCATIONS:
Overall Officials: Sara M Lippa, PhD, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Non-identified IPD will be made available through the Federal Interagency TBI Research (FITBIR) Database.
Time Frame: Data will be uploaded to the FITBIR system at the end of each funded year and at the completion of the study. This data will be made available to researchers using the FITBIR system 12 months after the end of the award period.
Access Criteria: FITBIR qualified investigators will be provided access.
URL: http://fitbir.nih.gov/